CLINICAL TRIAL: NCT03260933
Title: A Qualitative Study to Investigate Patients', Carers' and Providers' Perspectives on Integrated Care and Integrated Care Pathways for Frail Older People in Lambeth and Southwark, South London
Brief Title: Integrated Care for Frail Older People
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Euan Sadler, Senior Postdoctoral Research Fellow in Implementation Science, King's College London
Other Study IDs: IRAS Project ID: 226031
Record Dates: First submitted 2017-08-15; First posted 2017-08-24 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Frail Elderly Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention given. This is a qualitative interview study — This is a qualitative interview study

SUMMARY:
This is a qualitative interview study investigating patients', carers' and providers' perspectives on integrated care and integrated care pathways for frail older people in Lambeth and Southwark, south London.

ELIGIBILITY:
Inclusion Criteria:

1. Frail older people aged 65 years and over, including men and women with different levels of frailty.
2. Carers (family member, friend or neighbor) identified by the frail older participant as a main carer.
3. Health and social care professionals, care workers, service managers and commissioners working in different parts of the local health and care system (primary, secondary, community, social and voluntary care), reflecting a range of roles.

Exclusion Criteria:

1. Older people not identified as frail.
2. Frail older people who are unable to provide their informed consent to take part in the study, for example due to significant cognitive impairment.

Ages: 65 Years to 100 Years | Sex: All
Age Groups: Older Adult
Study Population: Frail older people, their carers and a range of providers.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Stakeholders perspectives as assessed by interview survey | Day 1
  Stakeholders perspectives as assessed by interview survey

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Euan Sadler, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No